CLINICAL TRIAL: NCT00480792
Title: Open-label, Randomized, and Multicentric Phase III Clinical Trial Comparing Three Strategies of Vaccination Against the Virus of Hepatitis B in HIV-1-infected Patients With CD4-positive T-lymphocytes Counts Above 200 permm3 ANRS HB 03 VIHVAC-B
Brief Title: Trial Comparing Three Strategies of Vaccination Against the Virus of Hepatitis B in HIV Infected Patients
Acronym: VIHVAC-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-003940-50; ANRS HB 03 VIHVAC-B
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: Hepatitis B vaccination; GenHevac-B Pasteur; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — GenHevac B Pasteur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): GenHevac-B 20 microgramme Intramuscular use at M0, M1, M6
  Interventions: Biological: GenHevac B Pasteur
- B (Experimental): GenHevac-B 40 microgramme Intramuscular use at M0, M1, M2, M6
  Interventions: Biological: GenHevac B Pasteur
- C (Experimental): GenHevac-B 4 microgramme Intradermal use at M0, M1, M2, M6
  Interventions: Biological: GenHevac B Pasteur

INTERVENTIONS:
Biological: GenHevac B Pasteur — Intra-muscular injection 20 microgramme Intramuscular use at M0, M1, M6
  Other Names: Sanofi Pasteur MSD
  Arms: A
Biological: GenHevac B Pasteur — Intra-muscular injection 40 microgramme intramuscular use at M0, M1,M2, M6
  Other Names: Sanofi Pasteur MSD
  Arms: B
Biological: GenHevac B Pasteur — GenHevac-B 4 microgramme Intradermal use at M0, M1, M2, M6
  Other Names: Sanofi Pasteur MSD
  Arms: C

SUMMARY:
In HIV infected patients, individuals exposed to the virus of Hepatitis B are more susceptible to develop a chronic and severe liver disease with a major risk of cirrhosis and liver cancer.

However, the existing protocol of vaccination against Hepatitis B is less efficient in HIV-infected patients than in non HIV-infected-patients, and, in case of response, its longevity has to be followed up carefully. This study compares the efficacy of the standard protocol vaccination with GenHevac-B and 2 other protocols, a double-dose of GenHevac-B and a set of intradermal injections of Genhevac-B, in HIV-infected patients with lymphocytes T CD4 level above 200 permm3.

DETAILED DESCRIPTION:
Comparison of 3 vaccination strategy against Hepatitis B in patients with HIV infection T CD4 above 200 per mm3

Intervention:

1. Arm A: GenHevac-B 20 microgramme Intramuscular use at M0, M1, M6
2. Arm B: GenHevac-B 40 microgramme Intramuscular use at M0, M1, M2, M6
3. Arm C: GenHevac-B 4 microgramme Intradermal use at M0, M1, M2, M6

ELIGIBILITY:
Inclusion Criteria:

Age Eligible for Study: 18 years - NA, Genders Eligible for Study: Both

Criteria

Inclusion criteria:

* HIV infection
* T CD4 count cell level above 200 per mm3
* Serology Hepatitis B negative (AgHBs, AbHBs and AbHBc negative)
* unchanged ARV for the last 3 months for patients who are receiving ARV at the screening visit
* Undetectable for the last 6 months with ARV for any patient with T CD4 level below 350 per mm3
* Pregnancy test negative at the screening and inclusion visits

Exclusion Criteria:

* Any injection of the vaccine against Hepatitis B in the medical history
* Acute cytolysis in the last 3 months with transaminases equal or above 5 times the upper normal range for HIV-HCV coinfected patients, or transaminases equal or above 2 times the upper normal for non coinfected patients
* Any vaccine received one month before the inclusion
* History of intolerance to any component of GenHevac-B
* Evolutive opportunistic infection treated the month before the screening visit
* Severe and acute pyretic infection or unexplained fever the week before inclusion
* Evolutive hemopathy or solid-organ cancer
* Prothrombin factor equal or below 50 percent and/or platelets equal or below 50 000 per mm3
* Immunosuppressive treatment or general corticotherapy (equal or above 0,5 mg per kg per day during above 7 days) in the last 6 months before the screening visit
* Previous Immunomodulating treatment (interferon, interleukin-2,etc) or plan in the next 6 months
* Splenectomy
* Decompensated cirrhosis (Child Pugh B or C)
* Kidney deficient function (creatinine clearance below 50 ml per mn)
* Other immunocompromised condition not related to HIV infection (solid-organ transplantation, chemotherapy in the last 6 months)
* Any participation to another clinical trial plan until Week 28

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
HIV-infected patients who seroconvert in the first two months after the last vaccination. Seroconversion is defined as antibodies AbHBs titers equal or above 10 mUI per ml. | two months after the last injection;week 28, month 18, month 30 and month 42

SECONDARY OUTCOMES:
According to the vaccine administration (IM or ID) comparison of AbHBs titers,permanence of the humoral response,intensity of clinical and biological events and predicting factors related to seroconversion | two months after the last injection; week 28, month 18, month 30 and month 42

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, Principal Investigator — CIC de vaccinologie Cochin-Pasteur 27, rue du Fb Saint Jacques 75014 Paris Fr; Fabrice Carrat, MD, Study Chair — Inserm U707 27, rue de Chaligny 75571 Paris cedex 12 Fr
Locations (1):
- Hopital Cochin CIC de vaccinologie, Paris, France

REFERENCES:
- [Derived] Launay O, Rosenberg AR, Rey D, Pouget N, Michel ML, Reynes J, Neau D, Raffi F, Piroth L, Carrat F; ANRS HB03 VIHVAC-B (Trial Comparing 3 Strategies of Vaccination Against the Virus of Hepatitis B in HIV-Infected Patients) Group. Long-term Immune Response to Hepatitis B Virus Vaccination Regimens in Adults With Human Immunodeficiency Virus 1: Secondary Analysis of a Randomized Clinical Trial. JAMA Intern Med. 2016 May 1;176(5):603-10. doi: 10.1001/jamainternmed.2016.0741. PMID 27064975
- [Derived] Launay O, van der Vliet D, Rosenberg AR, Michel ML, Piroth L, Rey D, Colin de Verdiere N, Slama L, Martin K, Lortholary O, Carrat F; ANRS HB03 VIHVAC-B Trial. Safety and immunogenicity of 4 intramuscular double doses and 4 intradermal low doses vs standard hepatitis B vaccine regimen in adults with HIV-1: a randomized controlled trial. JAMA. 2011 Apr 13;305(14):1432-40. doi: 10.1001/jama.2011.351. PMID 21486976